CLINICAL TRIAL: NCT03269864
Title: Use of Perforator Flaps for Leg and Foot Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Adel, Principal investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17200122
Record Dates: First submitted 2017-08-28; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Post Traumatic Skin Defect in Leg and Foot
MeSH Terms: interventions — Perforator Flap

STUDY DESIGN:
Intervention Model Description: two arms, one will be managed by pedicled perforator flaps the other will be managed by free perforator flaps
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pedicled perforator flaps (Active Comparator): Once the perforator is identified, the flap will be designed around the perforator or perforators according to the location and size of the defect.
  A tourniquet is inflated without prior exsanguination. This maneuver facilitates identification of perforators as they remain filled with the blood.
  An exploratory incision along the margin of flap is made keeping the position of marked perforator in mind. The incision is made through the skin, subcutaneous tissue, deep fascia (sub-fascial approach) and the perforator vessel is directly visualized. The incision is initially always made from one side of the flap only to properly identify the perforator.
  Careful and meticulous dissection is done in a blunt way isolating the perforator.
  After deflation of the tourniquet, hemostasis is performed.
  Interventions: Procedure: perforator flaps
- free perforator flaps (Active Comparator): A two-team approach is used for microvascular free tissue transfer. The first team starts exploring the limb for the recipient vessel. The second team simultaneously begins elevating the perforator flap and its vascular pedicle.
  Microvascular anastomosis will be carried out under operating microscope for one artery and one or two accompanying veins.
  Interventions: Procedure: perforator flaps

INTERVENTIONS:
Procedure: perforator flaps — 40 patients with post traumatic skin defect at leg and foot will be managed by perforator flaps, 20 with pedicled perforator flaps and other 20 with free perforator flaps

SUMMARY:
Perforator vessels are those where the source artery is deep and the branch that carries blood to the fasciocutaneous tissues passes through the overlying deep fascia.

Soft tissue defects in the lower extremity, especially distal third of leg, present a challenge to reconstructive surgeons due to lack of reliable local flaps, conventional reconstructive options include split skin grafting, local random fasciocutaneous flaps, cross leg fasciocutaneous flap, pedicled muscular or musculocutaneous flaps or microvascular free tissue transfer. All these procedures have their limitations and associated morbidity at donor site

DETAILED DESCRIPTION:
Taylor and Palmer defined an angiosome as a three-dimensional vascular territory supplied by a source artery and vein through branches for all tissue layers between the skin and the bone, and showed that between neighboring angiosomes there are choked and true anastomotic arteries.

Koshima and Soeda in 1989, described an inferior epigastric artery skin flap without the rectus abdominis muscle for reconstruction of floor of mouth, began the era of perforator flaps.

The big popularity gained by the local perforator flaps was due to their main advantages: 1) Sparing of the source artery and underlying muscle and fascia, 2) Combining the very good blood supply of a musculocutaneous flap with the reduced donor-site morbidity of a skin flap, 3) Replacing like with like, 4) Limiting the donor-site to the same area, 5) Possibility of completely or partially primarily closure, 6) Technically less demanding, because they are microsurgical procedures, but without microvascular sutures, 7) Shorter operating time.

ELIGIBILITY:
Inclusion Criteria:

1. Traumatic soft tissue defects on foot and leg.
2. Simple defects i.e., soft tissue loss, with or without, tendon injury.
3. Patients from 6 years to 60 years old

Exclusion Criteria:

1. Other causes of soft tissue defects e.g. (Diabetic, Vascular, post malignant resection).
2. Complex defects (soft tissue with bone injury).
3. Patients below 6 years or above 60 years old.
4. Patients with debilitating diseases e.g chronic renal failure, diabetes mellitus….etc.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-09-05 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the perforator flap | This will be assessed in the first week postoperative
  The perforator flap will be assessed regarding (color, temperature, capillary refilling, congestion, blistering).

IPD SHARING:
Plan to Share IPD: No